CLINICAL TRIAL: NCT01377883
Title: Clown Care for Botulinum Toxin (BTX)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Hilla Ben-Pazi, PI, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL_BTX2011
Record Dates: First submitted 2011-06-19; First posted 2011-06-22 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Cerebral Palsy; Pain
Keywords: Needle, Anxiety, Pain, Clowns
MeSH Terms: conditions — Cerebral Palsy; Pain; Anxiety Disorders

ARMS (2):
- Standard intervention (Sham Comparator): Preparation and information: the doctor and nurse explained the steps of the procedure: placing EMG electrodes, wiping the area with an alcohol swab, cooling with ethyl chloride, needle insertion into the muscle and the importance of EMG noise.
  Memory change and positive reinforcement: medical staff present spoke to the child positively and offered prizes, among which the child could choose.
  Volunteer attendance: as part of the control session, receiving no particular instructions in relation to the child's potential pain during the procedure.
  Interventions: Other: standard
- clown care (Experimental): Cognitive coping: encouraging a child to cope with the challenge. Imagery: a cognitive technique used to encourage the child to cope with the pain and distress of the procedure by imagining a pleasant object or experience Empowerment: the child is made to feel empowered by controlling the actions of the clown Reflecting emotions: the clown, sensing the state of the child, plays it out in an exaggerated fashion.
  Interventions: Behavioral: clown care

INTERVENTIONS:
Other: standard — Preparation and information regarding the BTX procedure: placing EMG electrodes, wiping the area with an alcohol swab, cooling with ethyl chloride, needle insertion into the muscle and the importance of EMG noise.
  Injection performed under EMG guidance. Two sites of injection per muscle were used to enhance diffusion. The child could often see the procedure when the upper limb was treated but not during lower limb injections.
  Memory change and positive reinforcement: Following the BTX injection, the medical staff present spoke to the child positively and offered prizes Volunteer attendance: In the daycare unit there are young volunteers routinely present, assisting with technical aspects of the procedure.
  Arms: Standard intervention
Behavioral: clown care — Cognitive coping Imagery Empowerment Reflecting emotions
  Arms: clown care

SUMMARY:
Children with cerebral palsy (CP) undergo multiple painful procedures such as Botulinum toxin (BTX) injections that are administered several times a year. While clown care reduces preoperative anxiety, its effect on painful procedures has not been assessed. We hypothesized that medical clowning reduces pain and anxiety during BTX injections.

DETAILED DESCRIPTION:
PATIENTS AND METHODS: Twenty five children with CP (mean age 7.4±4.8 years; 19 boys), enrolled in this randomized controlled study underwent BTX injections (3±1.7 muscles per procedure). Prior to treatment each child was assigned to receive either medical clown intervention (study) or standard care (control). Outcome measure was the Visual Analogue Scale (VAS) as reported by the child (n =14) or parent (n =11) prior and subsequent to each procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children with CP for whom BTX treatment was indicated

Exclusion Criteria:

* Children with minimal communication skills (n =1)
* Autistic spectrum disorders (n =1)
* Severe anxiety requiring general anesthesia (n =1)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | sevral minutes before and after BTX injections
  Visual Analogue Scale by the child before after BTX injection. Parent rated the pain if the child was younger than 5 years or cognitively impaired

REFERENCES:
- [Derived] Ben-Pazi H, Cohen A, Kroyzer N, Lotem-Ophir R, Shvili Y, Winter G, Deutsch L, Pollak Y. Clown-care reduces pain in children with cerebral palsy undergoing recurrent botulinum toxin injections- A quasi-randomized controlled crossover study. PLoS One. 2017 Apr 17;12(4):e0175028. doi: 10.1371/journal.pone.0175028. eCollection 2017. PMID 28414728